CLINICAL TRIAL: NCT01564043
Title: Internet Walking Program and Pedometer in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Boston Healthcare System (U.S. Federal Agency)
Collaborators: University of Michigan (Other); VA Ann Arbor Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Marilyn Moy, MD, VA Boston Healthcare System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VABHS2328
Record Dates: First submitted 2012-03-23; First posted 2012-03-27 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: COPD; Internet Access
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- website and pedometer (Experimental)
  Interventions: Behavioral: website and pedometer

INTERVENTIONS:
Behavioral: website and pedometer — use of pedometer and website

SUMMARY:
Higher levels of physical activity are associated with better functional status, fewer hospital admissions, and lower mortality. The investigators studied the feasibility and safety of a novel program that combines a pedometer with a website to increase walking. This is a pilot study.

ELIGIBILITY:
Inclusion Criteria:

* COPD
* able to ambulate
* internet access

Exclusion Criteria:

* current pulmonary rehab

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Daily step count | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- VABoston Healthcare System, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Moy ML, Weston NA, Wilson EJ, Hess ML, Richardson CR. A pilot study of an Internet walking program and pedometer in COPD. Respir Med. 2012 Sep;106(9):1342-50. doi: 10.1016/j.rmed.2012.06.013. Epub 2012 Jul 12. PMID 22795984